CLINICAL TRIAL: NCT07325227
Title: Remimazolam for Sedation in Cataract Surgery, A Phase IV, On-label, Blinded Study
Brief Title: Study of Remimazolam for Cataract Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fred E, Shapiro (Other)
Collaborators: Eagle Pharmaceuticals, Inc. (Industry); Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Sponsor-Investigator, Fred E, Shapiro, Principal Investigator, Massachusetts Eye and Ear Infirmary
Organization: Massachusetts Eye and Ear Infirmary (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2025P002034
Record Dates: First submitted 2025-12-09; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Cataract Surgery Anesthesia
Keywords: remimazolam; cataract surgery
MeSH Terms: interventions — remimazolam; Hypnotics and Sedatives

STUDY DESIGN:
Intervention Model Description: Subjects will be scheduled for cataract surgery in both eyes and they will serve as their own control, having sedation with the study drug remimazolam in one cataract surgery, and the standard of care sedation drug in the second surgery. To control for "second eye syndrome" a phenomenon where patients report increased discomfort, sensitivity, and / or slower healing at their second cataract surgery compared to the first, (even if no preoperative or intraoperative factor for that opinion could be identified) half of the subjects will have remimazolam as a sedative in their first cataract surgery and half will have it at the second surgery. Subjects will be blinded as to which sedation drug is used in each surgery.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 Cataract Surgery performed with remimazolam as sedative (Experimental): Subjects are serving as their own control. Subjects are scheduled for cataract surgery in both eyes. Sedation will be remimazolam in one eye and the standard of care in the other eye. The order of sedation will be randomly determined (50% of subjects will have remimazolam in the first eye surgery and 50% will have it in the second eye surgery.) Subjects will be blinded as to which sedation is provided at each surgery.
  Interventions: Drug: Arm 1 Cataract Surgery performed with remimazolam as sedative
- Arm 2 Cataract Surgery performed with a standard of care sedative (Placebo Comparator): Subjects are serving as their own control. Subjects are scheduled for cataract surgery in both eyes. Sedation in this arm will be the standard of care. The order of sedation will be randomly determined (50% of subjects will have remimazolam in the first eye surgery and 50% will have it in the second eye surgery.) Subjects will be blinded as to which sedation is provided at each surgery.
  Interventions: Drug: Arm 2 Cataract Surgery performed with standard of care sedative

INTERVENTIONS:
Drug: Arm 1 Cataract Surgery performed with remimazolam as sedative — Sedation will be remimazolam in one eye and the standard of care in the other eye.
  Arms: Arm 1 Cataract Surgery performed with remimazolam as sedative
Drug: Arm 2 Cataract Surgery performed with standard of care sedative — Standard of care sedative will be used during surgery.
  Arms: Arm 2 Cataract Surgery performed with a standard of care sedative

SUMMARY:
The goal of this clinical trial is to learn if the use of the sedative remimazolam improves the safety of patients having cataract surgery by decreasing the number of sedation-related complications during and after surgery, and shortening post-surgical cognitive recovery time.

DETAILED DESCRIPTION:
Remimazolam (Byfavo) is a novel benzodiazepine approved by the U.S. Food and Drug Administration in July 2020 for sedation in patients undergoing procedures less than 30 minutes in duration. Remimazolam is a rapid onset/offset benzodiazepine, designed to be rapidly metabolized without active metabolites reduce the changes in cognitive function known to occur after even a brief exposure to a sedative. This study will use remimazolam on-label to sedate patients having cataract surgeries that take less than 30 minutes to perform. The investigator is studying the use of remimazolam in cataract surgery because the investigator think it will improve patient safety by shortening post-surgery cognitive recovery time and decreasing the number of sedation-related complications.

ELIGIBILITY:
Inclusion Criteria:

* Subject is planning to have cataract surgery in both eyes
* The surgeon estimates that each cataract surgery are estimated to take less than 30 minutes
* Subject is aged 55 to 90 years old
* Surgeries will take place on the main campus of Mass Eye and Ear at 243 Charles St., Boston for at least the first year. In the future, surgeries may also occur at Mass Eye and Ear Longwood Surgical Ambulatory Care Center.
* Subject is able to understand the consent form and sign the consent
* ASA 1-3 (possible breakdown numbers of 5, 10, 10, 5)

Exclusion Criteria • Subject does not speak or read English

* Subject has a history of difficulty with sedation during procedures
* The surgeon estimates that one of the planned cataract surgeries is estimated to take longer than 30 minutes
* Subject uses concomitant home narcotic or anxiolytic
* Subject uses O2
* Subject has a history of cognitive decline
* A history of severe hepatic impairment

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
The number of sedation-related adverse events | Subjects consent to participate in study on day of surgery. AE data will be collected during surgery and through the following day when patient is contacted for follow-up. Adverse events will be documented up to one week after surgery should they occur
  The number of sedation-related adverse events from the time sedation is administered at the start of surgery through up to one week post-surgery.
The severity of sedation-related adverse events | Subjects consent to participate in study on day of surgery. AE data will be collected during surgery and through the following day when patient is contacted for follow-up. Adverse events will be documented up to one week after surgery should they occur
  The severity (mild, moderate or severe) of sedation-related adverse events
The duration of sedation-related adverse events | Subjects consent to participate in study on day of surgery. AE data will be collected during surgery and through the following day when patient is contacted for follow-up. Adverse events will be documented up to one week after surgery should they occur
  The duration, in minutes, hours, or days of sedation-related adverse events
Time that subject remains in the post anesthesia care unit (PACU) | Minutes starting with arrival in PACU after surgery until subject meets criteria for discharge
  Length of time in minutes that subject remains in the post anesthesia care unit (PACU) until he or she meets criteria for discharge. We are recruiting subjects whose cataract surgery is deemed uncomplicated and anticipated to last no more than 30 minutes. This is required to use remimazolam on label. We anticipate that subjects would be in the PACU for less than sixty minutes, but that the use of remimazolam will lead to discharge in less than 30 minutes.

SECONDARY OUTCOMES:
Subjects' scores using the Aldrete Postanesthetic Recovery assessment | During the time subject is in the post anesthesia care unit (PACU)
  Subjects' scores on repeated assessments made by staff while they are in the PACU using the Aldrete Postanesthetic Recovery Score system.
  The Aldrete Scoring System consists of 5 clinically relevant parameters reflecting physiological recovery from anesthesia: muscle activity, respiration, circulation, consciousness, and oxygenation. Each category is assigned a score of 0, 1, or 2, with a maximum possible total score of 10.
Subjects' scores on the Richmond Agitation Sedation Scale (RASS) | During the time subject is in the post anesthesia care unit (PACU)
  Subjects' scores on repeated assessments made by staff while they are in the PACU using the Richmond Agitation Sedation Scale (RASS).
  The Richmond Agitation Sedation Scale (RASS) was developed to assess the level of alertness and agitated behavior in patients who have received sedation. It is a 10-point scale ranging from -5 to +4. Levels -1 to -5 denote 5 levels of sedation and levels +1 to +4 describe increasing levels of agitation.
Subjects' scores on patient satisfaction questionnaires | Questionnaire will be completed the day after surgery
  Subjects will be asked to complete a questionnaire regarding their satisfaction with the sedation they received and their post-surgical recovery

OTHER OUTCOMES:
Patients' Indirect costs | 1 year
  We aim to compare subjects' indirect costs associated with post-surgical care i.e. time spent in the PACU prior to discharge post-surgery, and the time clinicians spend providing follow-up care related to the surgery in the weeks following discharge. We would like to compare standard of care vs. remimazolam.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Study results will be published in a medical journal.
Supporting Information: ICF, CSR
Time Frame: Study consent form will be added to this record after the documents are IRB approved. Data collection will be complete in 2027. Data will be analyzed in 2027 and the report will be published in 2028. We do not anticipate making the full data set available to others.
Access Criteria: The consent form will be available to members of the public that read this record on Clinicaltrials.gov.

REFERENCES:
- [Background] Alqudah A, Al-Dwairi R, Sharayah A, Al-Qudah NS, Almustafa YS, Al-Qudah A, Alharahsheh D, Al Awam RK, Al-Qudah H, Aleshawi A. Second Eye Syndrome: Patients' Perspectives Regarding First Eye versus Second Eye Phacoemulsification and Intraocular Lens Implantation Surgery. Patient Prefer Adherence. 2025 Jul 19;19:2081-2094. doi: 10.2147/PPA.S534166. eCollection 2025. PMID 40704218